CLINICAL TRIAL: NCT07369765
Title: Drug-Coated Balloon Versus Drug-eluting Stent Angioplasty for Treatment of Chronic Total Occlusion
Brief Title: Drug-Coated Balloon Versus Drug-eluting Stent Angioplasty for Treatment of Chronic Total Occlusion - The DCB-CTO Trial
Acronym: DCB-CTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Sevket Gorgulu, professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-BIAEK/12-9
Record Dates: First submitted 2026-01-03; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: CHRONIC TOTAL OCCLUSION; DRUG COATED BALLOON; CORONARY ARTERY DISEASE
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug Coated Balloon Group (Active Comparator): For this study, only one paclitaxel-coated balloon platform (Protégé™ Drug-Coated Balloon, Translumina, India) will be used in the drug-coated balloon group. The Protégé balloon catheter will be inflated for 1 minute in the chronic total occlusion segment. If multiple inflations are required with the same balloon, additional inflations of 30 seconds with an increase of 2 atm compared to the previous inflation will be allowed, up to a maximum of three inflations, which is a unique feature of the M3i DCB technology. The use of more than one drug-coated balloon is permitted if clinically required. All devices used are commercially available and used according to the manufacturer's instructions for use.
  Interventions: Device: Drug Coated Balloon Group
- Drug-Eluting Stent Group (Active Comparator): In the drug-eluting stent group, any commercially available CE-certified second-generation drug-eluting stent will be allowed for the treatment of chronic total occlusion. Stent implantation will be performed according to standard clinical practice and the manufacturer's instructions for use. The use of more than one drug-eluting stent is permitted if deemed necessary by the operator. All devices used in this study are commercially available, and the instructions for use can be found in the trial master file and investigator site file.
  Interventions: Device: Drug-Eluting Stent Group

INTERVENTIONS:
Device: Drug-Eluting Stent Group — In the drug-eluting stent group, any commercially available CE-certified second-generation drug-eluting stent will be allowed for the treatment of chronic total occlusion. Stent implantation will be performed according to standard clinical practice and the manufacturer's instructions for use. The use of more than one drug-eluting stent is permitted if deemed necessary by the operator. All devices used in this study are commercially available, and the instructions for use can be found in the trial master file and investigator site file.
  Arms: Drug-Eluting Stent Group
Device: Drug Coated Balloon Group — Percutaneous coronary intervention using a drug-coated balloon for the treatment of chronic total occlusion. The drug-coated balloon is used according to standard clinical practice and the manufacturer's instructions for use.
  Arms: Drug Coated Balloon Group

SUMMARY:
Chronic total occlusion (CTO) remains one of the most challenging lesions in coronary artery disease management. Percutaneous coronary intervention using drug-eluting stents is currently a standard treatment approach; however, drug-coated balloon angioplasty has emerged as a potential alternative strategy.

This study aims to compare the clinical and angiographic outcomes of drug-coated balloon angioplasty versus drug-eluting stent implantation in patients undergoing percutaneous coronary intervention for chronic total occlusion. The study will include adult patients diagnosed with CTO who meet the predefined eligibility criteria. Outcomes related to procedural success and follow-up results will be evaluated to assess the effectiveness of both treatment strategies.

DETAILED DESCRIPTION:
Chronic total occlusion (CTO) represents one of the most complex and technically demanding lesion subsets in the management of coronary artery disease. CTO lesions are characterized by complete coronary artery occlusion with Thrombolysis in Myocardial Infarction (TIMI) grade 0 flow for a duration of at least three months and are frequently associated with increased procedural complexity, longer intervention times, and higher rates of restenosis and repeat revascularization.

Percutaneous coronary intervention (PCI) with drug-eluting stent (DES) implantation is currently considered the standard interventional treatment for CTO lesions and has demonstrated favorable outcomes in terms of vessel patency and symptom relief. Nevertheless, DES implantation is associated with potential limitations, including permanent metallic implantation, risk of late stent failure, in-stent restenosis, and the need for prolonged dual antiplatelet therapy. As a result, alternative strategies that avoid permanent implants have gained increasing interest.

Drug-coated balloon (DCB) angioplasty has emerged as a promising alternative approach in selected coronary lesions by delivering antiproliferative drugs to the vessel wall without leaving behind a permanent scaffold. The use of DCBs may offer theoretical advantages in CTO interventions, including preservation of native vessel anatomy, reduced risk of late adverse events, and potential facilitation of future interventions if needed. However, evidence directly comparing DCB angioplasty with DES implantation in the setting of CTO remains limited.

The present study is designed to compare the clinical and angiographic outcomes of DCB angioplasty versus DES implantation in adult patients undergoing PCI for chronic total occlusion. Eligible patients with a confirmed diagnosis of CTO who meet predefined inclusion and exclusion criteria will be enrolled. The choice of revascularization strategy will follow the study protocol, and procedural success will be assessed according to standardized angiographic and clinical definitions.

Clinical outcomes, including procedural success, major adverse cardiovascular events, need for repeat revascularization, and other relevant follow-up parameters, will be evaluated during the follow-up period. Angiographic outcomes, such as vessel patency and restenosis, will also be assessed when applicable. By comparing these two treatment strategies, this study aims to provide further evidence to inform optimal interventional management of CTO lesions and to clarify the potential role of drug-coated balloon angioplasty as an alternative to drug-eluting stent implantation in this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

* • Definite or probable CTO as per CTO-ARC definition

  * CTO length ≥ 20 mm and ≤ 40 mm;
  * High likelihood (≥90 %) of CTO-PCI success (balance between CTO lesion complexity and operator expertise);
  * Successful treatment of any non-CTO lesions at least 1 month before randomization;
  * CTO lesion location in a vessel segment with diameter ≥ 2.5 mm;
  * Successful intraplaque (intraluminal) wiring (extraplaque tracking < 10 mm or < 50% of occlusion length) with no flow-limiting dissection and a TIMI flow ≥ 2 after initial predilation with NC balloon.

Exclusion Criteria:

* Life expectancy < 1 year as result of non-cardiac conditions;
* Multiple CTO lesions that require recanalization;
* Target lesion is an in-stent CTO;
* Angiographic grade 3 calcifications in the CTO segment (Appendix 2);
* Recent acute coronary syndrome (< 1 month);
* Cardiogenic shock or inability to stay in supine position for long time;
* Severe kidney failure (eGFR ≤ 30 mL/min);
* Any planned non-CTO PCI < 12 months after randomization;
* Anticipated less compliance of the patients to complete the following or taking medical therapy;
* Patient or legal representative unable or unwilling to provide written informed consent prior to study enrollment;
* Pregnancy or childbearing age unless a recent pregnancy test is negative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Target vessel patency evaluated by QCA | From enrollment to the 6th month angiograhic follow-up
  Angiographic patency of the treated CTO vessel
Major adverse cardiovascular events (MACE) | From the enrollment to the end of 6th month follow-up
  Composite of cardiac death, myocardial infarction, and target vessel revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided